CLINICAL TRIAL: NCT01773070
Title: A Follow-up Study to Assess Resistance and Durability of Response to AbbVie Direct-Acting Antiviral Agent (DAA) Therapy in Subjects Who Participated in Phase 2 or 3 Clinical Studies for the Treatment of Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Follow up Study Designed to Obtain Long Term Data on Participants Who Either Achieved a Sustained Virologic Response or Did Not Achieve a Sustained Virologic Response in an AbbVie Sponsored Hepatitis C Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M13-102; 2012-003073-26 (EudraCT Number)
Record Dates: First submitted 2012-11-19; First posted 2013-01-23 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Hepatitis C virus; Direct Acting Antiviral; Sustained Virologic Response; Hepatitis C; Persistence of treatment-emergent substitutions
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — paritaprevir; dasabuvir; ombitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Other): Participants who received ABT-450, ABT-333 or ABT-267 at any dose level in an eligible prior AbbVie Phase 2 or 3 study for the treatment of chronic HCV, followed for up to 3 years post-treatment.
  Interventions: Drug: ABT-450/ritonavir; Drug: ABT-333; Drug: ABT-267

INTERVENTIONS:
Drug: ABT-450/ritonavir — ABT-450 coformulated with ritonavir. Drug is not administered -- this study is follow-up for participants previously receiving the drug.
  Other Names: ABT-450 also known as paritaprevir
Drug: ABT-333 — Drug is not administered -- this study is follow-up for participants previously receiving the drug.
  Other Names: dasabuvir
Drug: ABT-267 — Drug is not administered -- this study is follow-up for participants previously receiving the drug.
  Other Names: ombitasvir

SUMMARY:
A follow-up study to assess resistance and durability of response to 3 experimental drugs ABT-450/r, ABT-267, and ABT-333 in participants who have participated in AbbVie Phase 2 or 3 clinical studies with these agents for the treatment of chronic hepatitis C virus (HCV). Studies include: M11-646 (NCT01716585), M11-652 (NCT01464827), M12-746 (NCT01306617), M12-998 (NCT01458535), M13-098 (NCT01715415), M13-099 (NCT01704755), M13-386 (NCT01563536), M13-389 (NCT01674725)' M13-393 (NCT01685203), M13-961 (NCT01767116), M14-002 (NCT01833533), and M14-103 (NCT01911845).

ELIGIBILITY:
Inclusion Criteria:

* Subject has received at least one dose of ABT-450, ABT-333 or ABT-267 in a prior AbbVie HCV Phase 2 or 3 study which is being submitted as a US IND.
* The interval between the last dose of the AbbVie DAA therapy from the previous clinical study and enrollment in Study M13-102 must be no longer than 2 years.
* The subject must voluntarily sign and date the informed consent form.
* Subject completed the post-treatment period of an eligible prior study.

Exclusion Criteria:

* The investigator considers the subject unsuitable for the study for any reasons.
* Receipt of any investigational product from Day 1 and while enrolled in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2013-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This follow-up study was open to participants from AbbVie studies M11-646 (NCT01716585), M11-652 (NCT01464827), M12-746 (NCT01306617), M12-998 (NCT01458535), M13-098 (NCT01715415), M13-099 (NCT01704755), M13-386 (NCT01563536), M13-389 (NCT01674725)' M13-393 (NCT01685203), M13-961 (NCT01767116), M14-002 (NCT01833533), and M14-103 (NCT01911845).
Groups:
- All Participants: Participants who received ABT-450, ABT-333 or ABT-267 at any dose level in an eligible prior AbbVie Phase 2 or 3 study for the treatment of chronic hepatitis C virus (HCV), followed for up to 3 years post-treatment.
Period: Overall Study
Arm/Group | All Participants
Started | 478
Completed | 397
Not Completed | 81
Not completed — Withdrawal by Subject | 24
Not completed — Lost to Follow-up | 39
Not completed — Other | 15
Not completed — Death (unrelated to study procedures) | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 478
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227
  Male | 251

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Relapse12overall With and Without New HCV Infection
Description: Relapse is defined as a confirmed HCV ribonucleic acid (RNA) ≥ the lower limit of quantitation (LLOQ) at any time during the post-treatment period for a participant who had HCV RNA < LLOQ at the end of treatment. Relapse12overall is defined as a confirmed HCV RNA ≥ LLOQ at any time after the sustained virologic response at Week 12 post-dosing (SVR12) assessment time point for a participant who achieved SVR12 and had post-SVR12 HCV RNA data available. SVR12 is defined as HCV RNA < LLOQ in the SVR12 window (12 weeks after the last actual dose of study drug) without any confirmed quantifiable (≥ LLOQ) post-treatment value before or during that SVR window. New HCV infection is defined as re-infection with a different HCV isolate.
Time Frame: Up to 3 years post-treatment
Population: Participants who achieved SVR12 and had post-SVR12 HCV RNA data available. Participants who did not have any post-treatment HCV RNA values were excluded from the relapse analyses.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 457
percentage of participants
  Relapse12overall With New HCV Infection | 0.2
  Relapse12overall Without New HCV Infection | 0.2

2. Primary Outcome: Number of HCV Genotype (GT)1a-Infected Participants With Persistence of Treatment-Emergent Substitutions in NS3, NS5A, or NS5B
Description: The persistence of specific hepatitis C amino acid variants (treatment-emergent substitutions) associated with drug resistance in NS3, NS5A, or NS5B was evaluated in participants who had not achieved SVR12. Post-baseline time points were calculated relative to the last dose of study drug in the previous study.
Time Frame: from the last dose of study drug in the previous study up to 3 years post-treatment
Population: GT1a-infected participants who experienced virologic failure after receiving ABT-450, ABT-333 or ABT-267, and had not achieved SVR12 and had post-baseline sequencing data for NS3, NS5A, or NS5B at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 18
Participants
  NS3: time of failure | 7
  NS3: post-treatment week 48: number analyzed (Participants) | 7
  NS3: post-treatment week 48 | 0
  NS5A: time of failure | 13
  NS5A: post-treatment week 48: number analyzed (Participants) | 10
  NS5A: post-treatment week 48 | 10
  NS5A: post-treatment week 96: number analyzed (Participants) | 8
  NS5A: post-treatment week 96 | 6
  NS5A: post-treatment week 132: number analyzed (Participants) | 8
  NS5A: post-treatment week 132 | 4
  NS5B: time of failure: number analyzed (Participants) | 15
  NS5B: time of failure | 7
  NS5B: post-treatment week 24: number analyzed (Participants) | 4
  NS5B: post-treatment week 24 | 3
  NS5B: post-treatment week 96: number analyzed (Participants) | 5
  NS5B: post-treatment week 96 | 1

3. Secondary Outcome: Percentage of Participants Who Experienced Relapse12 Without and With New HCV Infection
Description: Relapse is defined as a confirmed HCV RNA ≥ LLOQ at any time during the post-treatment period for a participant who had HCV RNA < LLOQ at the end of treatment. Relapse12 is defined as a confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after last actual dose of study drug (up to and including the SVR12 assessment time point) for a participant with HCV RNA < LLOQ at Final Treatment Visit who completed treatment.
Time Frame: From the end of treatment through 12 weeks post-treatment
Population: Participants with HCV RNA < LLOQ at Final Treatment Visit who completed treatment. Participants who did not have any post-treatment HCV RNA values were excluded from the relapse analyses.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 458
percentage of participants
  Relapse12 Without New HCV Infection | 2.0
  Relapse12 With New HCV Infection | 0

4. Secondary Outcome: Percentage of Participants Who Experienced Relapse24 Without and With New HCV Infection
Description: Relapse is defined as a confirmed HCV RNA ≥ LLOQ at any time during the post-treatment period for a participant who had HCV RNA < LLOQ at the end of treatment. Relapse24 is defined as a confirmed HCV RNA ≥ LLOQ within the sustained virologic response at Week 24 post-dosing (SVR24) window for a participant who achieved SVR12 and had HCV RNA data available in the SVR24 window.
Time Frame: From the end of treatment through 24 weeks post-treatment
Population: Participants who achieved SVR12 and had HCV RNA data available in the SVR24 window. Participants who did not have any post-treatment HCV RNA values were excluded from the relapse analyses.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 403
percentage of participants
  Relapse24 Without New HCV Infection | 0.2
  Relapse24 With New HCV Infection | 0

5. Secondary Outcome: Percentage of Participants Who Experienced Relapse˅Overall Without and With New HCV Infection
Description: Relapse is defined as a confirmed HCV RNA ≥ LLOQ at any time during the post-treatment period for a participant who had HCV RNA < LLOQ at the end of treatment. Relapse˅overall was defined as a confirmed HCV RNA ≥ LLOQ between end of treatment and up to and including the last HCV RNA measurement collected in the post-treatment Period for a participant with HCV RNA < LLOQ at Final Treatment Visit who completed treatment.
Time Frame: Up to 3 years post-treatment
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 458
percentage of participants
  Relapse˅overall Without New HCV Infection | 2.2
  Relapse˅overall With New HCV Infection | 0.2

ADVERSE EVENTS:
Time Frame: From last dose of direct-acting antiviral agent treatment in the previous study to last HCV RNA assessment in M13-102 (mean [SD] duration: 146.3 [28.16] weeks).
Description: Per protocol, only serious adverse events that the investigator considered to be causally related to study procedures (i.e., venipunctures) were collected in this study. Non-serious adverse events were not collected.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 3/478
Serious Adverse Events (participants affected / at risk) | 0/478
Other Adverse Events (participants affected / at risk) | 0/478

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.